CLINICAL TRIAL: NCT06706375
Title: A Comparison of Reversed-Ultrasound-Guided Dorsal Penile Nerve Block (RUS-DPBP) and DPNB in Circumcisions for Pediatric Patients
Brief Title: Compared Reversed US-Guided Dorsal Penile Nerve Block (RUSDPNB) with DPNB in Circumcisions for Pediatric Patients
Acronym: CIRCUSPRO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Patrick Schoettker, Professeur Patrick Schoettker, head of anesthesiology service, CHUV, Lausanne, Switzerland, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024-00420
Record Dates: First submitted 2024-11-20; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Circumcision; Ultrasound; Opioid Consumption; Penile Surgery
Keywords: circumcision; reversed ultrasound guided dorsal penile nerve block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- interventional (Experimental): Dorsal penile nerve block using ultrasound
  Interventions: Procedure: Using ultrasound for penile nerve block
- Control (Active Comparator): Dorsal penile nerve block using anatomical landmarks
  Interventions: Procedure: Dorsal Penile Block Anesthesia using landmarks

INTERVENTIONS:
Procedure: Using ultrasound for penile nerve block — 30% of men over the age of fifteen worldwide have had a circumcision according to a World Health Organization report. (1) This operation is common and should not be trivialized. A certain number of surgical complications should be considered, including pain, infections, excessive bleeding or hematomas. (1,2) Today, the use of opioids as intra- and postoperative analgesics in pediatric urological surgery remains predominant (3) but is the subject of increasing controversies. Indeed, the recent opioid crisis challenges us about their use and highlights their multiple side effects. First of all, their use involves significant risks, (4) including opioid-induced hyperalgesia and potential long-term effects. An increase in pain sensitivity within the 24 postoperative hours being proportional to intraoperative administration of high doses of opioids can be observed. (5) Long-term addiction is also questioned. Then, opioids don't appear to be the most effective per- and postoperative analgesi
  Arms: interventional
Procedure: Dorsal Penile Block Anesthesia using landmarks — Dorsal penile nerve block (DPNB) is LRA technique of choice for circumcisions and aims to anesthetize both dorsal penile nerves. (10-12) The name DPNB is used for blocks performed by determining precise dorsal anatomical landmarks and doing two distinct injections.
  Arms: Control

SUMMARY:
Circumcision is a widely performed surgical procedure. For this reason, optimal analgesic management is essential. Loco-regional anesthesia, particularly penile blocks, combined with general anesthesia is the technique of choice for managing analgesia during circumcisions.

Ultrasound is increasingly used in locoregional anesthesia techniques. There is already human research on penile blocks and the use of ultrasound. Studies carried out to date describe an optimization of pain relief in children after circumcision compared with the alternative technique without ultrasound, as well as a reduction in local complications due to injection. However, other studies tend to contradict these findings.

In order to provide additional knowledge and to verify whether ultrasound could provide you with more optimal relief after your circumcision, we are carrying out this study.

We are proposing to every patient aged 0 to under 18 who is going to undergo circumcision to take part in this project. A letter is sent to all potential participants no later than 3 days before the operation. We then discuss the matter in person during the pre-anaesthetic visit, which takes place by telephone or face-to-face no later than the day before the operation. Consent can be signed no later than the day of the operation. The cooling-off period is the same regardless of age.

Taking part in the study does not affect your operation in any way. On the day of the operation, you must report to the CHUV admissions desk. You will meet the anaesthetists on the day of the operation, who will again give you details of the anaesthesia and analgesic block. The block will take place in the operating room, prior to surgery.

In our study, participants are randomized into groups. This method is important for obtaining reliable results.

* Group 1 (intervention group): The penile block will be performed using ultrasound.
* Group 2 (control group): The penile block will be performed using anatomical landmarks.

This is a "single-blind" study, which means that only the anaesthetists, investigators and operating room team will be aware of the allocation to one of the two groups.

We will follow the participants and collect data on their opiate consumption; the different durations preoperatively, intraoperatively, postoperatively, back in the recovery room and before returning home; any complications as well as pain assessment.

DETAILED DESCRIPTION:
30% of men over the age of fifteen worldwide have had a circumcision according to a World Health Organization report. This operation is common and should not be trivialized. A certain number of surgical complications should be considered, including pain, infections, excessive bleeding or hematomas. Today, the use of opioids as intra- and postoperative analgesics in pediatric urological surgery remains predominant but is the subject of increasing controversies. Indeed, the recent opioid crisis challenges us about their use and highlights their multiple side effects. First of all, their use involves significant risks, including opioid-induced hyperalgesia and potential long-term effects. An increase in pain sensitivity within the 24 postoperative hours being proportional to intraoperative administration of high doses of opioids can be observed. Long-term addiction is also questioned. Then, opioids don't appear to be the most effective per- and postoperative analgesic drug. Its prescription could and should be reduced. In sum, a safe and effective anesthesia is paramount. Use of loco-regional anesthesia (LRA) during pediatric urological surgeries complements general anesthesia and thus offers more optimal postoperative analgesia.

Dorsal penile nerve block (DPNB) is LRA technique of choice for circumcisions and aims to anesthetize both dorsal penile nerves. The name DPNB is used for blocks performed by determining precise dorsal anatomical landmarks and doing two distinct injections. The main complications observed are lesions of the urethra, vascular complications (bleeding from the prepuce; hematomas) and failure of the block. In recent years, Ultrasound (US), a non-irradiating imaging technique widely used in LRA, has been used more and more to perform the DPNB and the procedure is well known and described. A decrease of the amount of opioid analgesics intraoperatively and postoperatively is observed when US is used. Postoperative pain scores are also better. Two methods of DPNB using US exist. In both approaches, probe is placed along the transverse plan. In the first one at the base of penis, with ventral visualization of structures, US-DPNB. In the second method, Reversed Ultrasound-Guided DPNB (RUS-DPNB), the penis is slightly retracted with probe placed dorsally, under the base of penis and above the scrotum. RUS-DPNB method will be used in this study. However, DPNB and RUS-DPNB are well described and used equally in daily practice.

The aim of this prospective study is to compare DPNB and RUS-DPNB in terms of efficacy, using cumulative analgesic dosage in morphine equivalent per kilogram. In the standard practice, the two methods are performed at discretion of every anaesthesiologist at CHUV. In fact, although RUS-DPNB is part of everyday practice at CHUV, it hasn't become the standard method, as the literature has a lack of data to prove its advantage over the standard method, DPNB.

ELIGIBILITY:
Inclusion Criteria:

* male
* undergoing circumcision
* informed consent

Exclusion Criteria:

* other surgery than circumcision in the same time
* contraindication to local anesthesia
* allergy to bupivacaine
* chronic opiates treatment

Max Age: 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — males only as it is circumcision
Enrollment: 216 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Total morphine equivalent | from enrollment to discharge from hospital, maximum 1 day
  total morphine equivalent will be cumulated and reported

SECONDARY OUTCOMES:
times | from enrollment to discharge from hospital, maximum 1 day
  - Anesthesia time, surgery time, total time in operating room, time in recovery room, time before discharge home
Adverse events | from enrollment to discharge from hospital, maximum 1 day
  - Incidence of adverse events of special interest (complications such as urine retention, bleeding and hematoma, nausea and vomiting).
Pain score using FLACC or FACES or VAS, from 0 (no pain) to 10 (worse pain) | from enrollment to discharge from hospital, maximum 1 day
  Maximal pain score measured and reported

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Beginning 1 year after publication with no end date
Access Criteria: Any researcher or journal contacting the PI with clear and well-founded request

REFERENCES:
- [Background] O'Sullivan MJ, Mislovic B, Alexander E. Dorsal penile nerve block for male pediatric circumcision--randomized comparison of ultrasound-guided vs anatomical landmark technique. Paediatr Anaesth. 2011 Dec;21(12):1214-8. doi: 10.1111/j.1460-9592.2011.03722.x. PMID 22023417
- [Background] Kirya C, Werthmann MW Jr. Neonatal circumcision and penile dorsal nerve block--a painless procedure. J Pediatr. 1978 Jun;92(6):998-1000. doi: 10.1016/s0022-3476(78)80386-2. PMID 660375
- [Background] Osmani F, Ferrer F, Barnett NR. Regional anesthesia for ambulatory pediatric penoscrotal procedures. J Pediatr Urol. 2021 Dec;17(6):836-844. doi: 10.1016/j.jpurol.2021.07.017. Epub 2021 Jul 24. PMID 34400101
- [Background] Carolan AMC, Parker KM, Grimsby GM. Opioid Use after Pediatric Urologic Surgery: Is It Really Needed? Urology. 2021 Dec;158:184-188. doi: 10.1016/j.urology.2021.04.012. Epub 2021 Apr 24. PMID 33901533